CLINICAL TRIAL: NCT02882581
Title: Metformin in Breast Cancer, Visualized With Positron Emission Tomography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Elias Immanuel Ordell Sundelin, MD, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-000132-18
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Metformin; Pharmacokinetics; Organic cation transporter; Multidrug and toxin extrusion; Pharmacogenetics; positron emission tomography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 11C-metformin uptake in breast cancer. Single center, single dose, open-label.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 11C-metformin (Experimental): All participants allocated to the study will be included in this arm
  Interventions: Radiation: 11C-metformin

INTERVENTIONS:
Radiation: 11C-metformin — 400MBq of 11C-metformin is injected in the cubital vein. The participant is then scanned for 120 min using Position Emission Tomography.

SUMMARY:
The general purpose of the trial is to investigate whether metformin is taken up into the breast tumor. Studies in the last few years have shown an effect of metformin on cell proliferation on breast cancer. It is though unclear whether the effect on tumor is direct, indirect or a combination of the two. The investigators plan to:

* investigate if metformin is taken up in breast cancer using our novel 11C-metformin tracer and positron emission tomography (PET)
* investigate whether the uptake is correlated to the amounts of organic cation transporters (OCT1-3, MATE 1 &2 and PMAT) using quantitive polymerase chain reaction (qPCR).

ELIGIBILITY:
Inclusion Criteria:

* over 50 years
* C. mammae
* Tumor size: > 10 mm in diameter
* Unilateral cancer
* WHO performance status 0-1

Exclusion Criteria:

* Severe heart- or kidney failure
* Pregnant or breast feeding
* If the patient is found not eligible for participation in the study på principal investigator

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Metformin uptake in breast cancer | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jessen, Prof,MD,PhD, Study Director — Department of Clinical Pharmacology, Aarhus University Hospital; Elias IO Sundelin, MD, Principal Investigator — Department of Clinical Medicine, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Nuclear Medicine & PET-center, Aarhus University Hospital, Aarhus
  - Department of Surgery, Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No